CLINICAL TRIAL: NCT00502034
Title: Adjuvant Low-dose Interleukin-2 (IL2) Plus Interferone-alpha (IFN) in Operable Renal Cell Cancer (RCC). Phase III, Randomized, Multicenter Trial of the Italian Oncology Group for Clinical Research (GOIRC).
Brief Title: Low-dose IL-2 Plus IFN-alpha Immunotherapy as Adjuvant Treatment of Renal Carcinoma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POLAR 01
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Carcinoma, Renal Cell
Keywords: Carcinoma, Renal Cell; Low-dose Interleukin; Adjuvant Immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interferon alpha-2; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-immunotherapy (Experimental): Immunotherapy with interferon-alpha and interleukin
  Interventions: Drug: Interferon Alfa-2a; Drug: Interleukin-2
- B-follow-up (No Intervention): Wait-and-see

INTERVENTIONS:
Drug: Interferon Alfa-2a — Interferon Alfa-2a in combination with Interleukin
  Arms: A-immunotherapy
Drug: Interleukin-2 — Interferon Alfa-2a in combination with Interleukin
  Arms: A-immunotherapy

SUMMARY:
The aim of this study is to compare the efficacy (in terms of event-free survival and overall survival) of an adjuvant therapy with IFN-alpha plus low-dose of IL2 vs a wait-and-see program in patient with radically operated renal cell carcinoma.

DETAILED DESCRIPTION:
For pts with non-metastatic RCC, no standard adjuvant treatment exists. Immunotherapy (IT) using IFN and/or IL2 is effective in metastatic disease setting. Low and chronically repeated doses of IL2 plus IFN induce a persistent stimulation of the immune system with no relevant toxicity.

Surgically treated RCC pts were randomized to the following arms: A) low-dose IT; B) control arm. IT consisted of a 4-week cycle of s.c. IL2 (5 days/wk, 1 million UI/sqm bid d 1,2 and 1 million UI/sqm x 1 d 3,4,5) + IFN (1,8 million UI/sqm d 3,5 of each week). Cycles were repeated every 4 months for the first 2 years and every 6 months for the remaining 3 years. Each patient received 12 cycles in 5 years. Inclusion criteria were as follows: histological diagnosis of RCC, age <75 yrs, radical or partial nephrectomy within the past 3 months, pT1 (diameter of T > 2,5 cm), T2, T3 a-b-c; pN0-pN3, M0; good cardiac and renal function and no autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis histologically confirmed of renal cells carcinoma (every histotype);
* Age < 75 years
* Radical surgical removal of the tumor: total or partial nephrectomy within previous 3 months
* Patient classified as T1 (with diameter > 2,5 cm), T2, T3 a-b-c; In presence of involvement of loco-regional lymph-nodes (staging N1, N2, N3, TNM class.), metastases should have been completely removed during nephrectomy
* Absence of distant metastases;
* Written informed consent

Exclusion Criteria:

* Tumor diameter equal or less than 2,5 cm;
* Previous chemotherapy or ormonotherapy o immunotherapy;
* Renal insufficiency >3 mg/dl);
* No symptomatic arrhythmias or autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 1994-07; Primary Completion 2007-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival: loco-regional, adrenal, kidney and distant-metastases were the events considered for event-free survival.

SECONDARY OUTCOMES:
Tolerability, toxicity and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Passalacqua, Medicine, Study Chair — Gruppo Oncologico Italiano di Ricerca Clinica; Carlo Buzio, Medicine, Study Chair — Parma University
Locations (8):
- Italy (8):
  - Carpi Hospital, Carpi, Modena
  - Ospedali Riuniti di Bergamo, Bergamo
  - Istituti Ospitalieri di Cremona, Cremona
  - Modena University Hospital, Modena
  - Parma University Hospital, Parma
  - Pavia University Hospital, Pavia
  - Ospedale "Guglielmo da Saliceto", Piacenza
  - Arcispedale Santa Maria Nuova, Reggio Emilia

REFERENCES:
- [Background] Passalacqua R, Buti S, Tomasello G, Longarini R, Brighenti M, Dalla Chiesa M. Immunotherapy options in metastatic renal cell cancer: where we are and where we are going. Expert Rev Anticancer Ther. 2006 Oct;6(10):1459-72. doi: 10.1586/14737140.6.10.1459. PMID 17069530
- [Background] Giacosa R, Santi R, Vaglio A, Pavone L, Ferrozzi F, Passalacqua R, Buzio C. "Late" regressions of metastases from renal cancer after a period of disease progression continuing the same intermittent low dose immunotherapy regimen. Acta Biomed. 2004 Aug;75(2):126-30. PMID 15481703
- [Background] Buzio C, Andrulli S, Santi R, Pavone L, Passalacqua R, Potenzoni D, Ferrozzi F, Giacosa R, Vaglio A. Long-term immunotherapy with low-dose interleukin-2 and interferon-alpha in the treatment of patients with advanced renal cell carcinoma. Cancer. 2001 Nov 1;92(9):2286-96. doi: 10.1002/1097-0142(20011101)92:93.0.co;2-i. PMID 11745283
- [Background] Buzio C, De Palma G, Passalacqua R, Potenzoni D, Ferrozzi F, Cattabiani MA, Manenti L, Borghetti A. Effectiveness of very low doses of immunotherapy in advanced renal cell cancer. Br J Cancer. 1997;76(4):541-4. doi: 10.1038/bjc.1997.422. PMID 9275034
- [Derived] Passalacqua R, Caminiti C, Buti S, Porta C, Camisa R, Braglia L, Tomasello G, Vaglio A, Labianca R, Rondini E, Sabbatini R, Nastasi G, Artioli F, Prati A, Potenzoni M, Pezzuolo D, Oliva E, Alberici F, Buzio C; POLAR-01 Trial Investigators. Adjuvant low-dose interleukin-2 (IL-2) plus interferon-alpha (IFN-alpha) in operable renal cell carcinoma (RCC): a phase III, randomized, multicentre trial of the Italian Oncology Group for Clinical Research (GOIRC). J Immunother. 2014 Nov-Dec;37(9):440-7. doi: 10.1097/CJI.0000000000000055. PMID 25304727